CLINICAL TRIAL: NCT04401319
Title: Repetitive Transcranial Magnetic Stimulation and Electroencephalography in Patients With Disorders of Consciousness
Brief Title: rTMS and EEG in DOC Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Liege (Other)
Collaborators: Therapiezentrum Burgau (Other)
Responsible Party: Principal Investigator, Olivia Gosseries, Principal Investigator, University of Liege
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: B0201941888
Record Dates: First submitted 2020-05-03; First posted 2020-05-26 (Actual); Last update posted 2023-12-12 (Actual); Status verified 2023-06

CONDITIONS: Disorder of Consciousness
Keywords: disorders of consciousness; transcranial magnetic stimulation
MeSH Terms: conditions — Consciousness Disorders | interventions — Cross-Over Studies

STUDY DESIGN:
Intervention Model Description: We will perform a 3 arm crossover trial. Subsequently, we will perform a longer protocol using a 3 arm parallel design.
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Sham Stimulation Group for Crossover Study (DLPFC + AG) (Sham Comparator): Sham stimulation will be delivered on the dorsolateral prefrontal cortex (DLPFC) and on the angular cortex (AG) using a sham coil in the crossover study.
  Interventions: Device: Sham Stimulation for Crossover Study
- DLPFC Stimulation Group for Crossover Study (Active Comparator): Real stimulation will be delivered on the left dorsolateral prefrontal cortex (DLPFC) using a real coil in the crossover study.
  Interventions: Device: DLPFC Stimulation for Crossover Study
- AG Stimulation Group for Crossover Study (Active Comparator): Real stimulation will be delivered on the left angular cortex (AG) using a real coil in the crossover study.
  Interventions: Device: AG Stimulation for Crossover Study
- Sham Stimulation Group for Parallel Study (DLPFC + AG) (Sham Comparator): Sham stimulation will be delivered on the dorsolateral prefrontal cortex (DLPFC) or on the angular cortex (AG) using a sham coil in the parallel study.
  Interventions: Device: Sham Stimulation for Parallel Study
- DLPFC Stimulation Group for Parallel Study (Active Comparator): Real stimulation will be delivered on the left dorsolateral prefrontal cortex (DLPFC) using a real coil in the parallel study.
  Interventions: Device: DLPFC Stimulation for Parallel Study
- AG Stimulation Group for Parallel Study (Active Comparator): Real stimulation will be delivered on the left angular cortex (AG) using a real coil in the parallel study.
  Interventions: Device: AG Stimulation for Parallel Study

INTERVENTIONS:
Device: Sham Stimulation for Crossover Study — Stimulation will be delivered on the dorsolateral prefrontal cortex (DLPFC) or the angular cortex (AG) using a sham coil for 20 minutes with a frequency of 20Hz (train duration: 4s; inter-train interval: 26s; 3200 pulses at 80% of the resting motor threshold ) in one session. A single session will be conducted.
  Arms: Sham Stimulation Group for Crossover Study (DLPFC + AG)
Device: DLPFC Stimulation for Crossover Study — Stimulation will be delivered on the left dorsolateral prefrontal cortex (DLPFC) using a real coil for 20 minutes with a frequency of 20Hz (train duration: 4s; inter-train interval: 26s; 3200 pulses at 80% of the resting motor threshold ) in one session. A single session will be conducted.
  Arms: DLPFC Stimulation Group for Crossover Study
Device: AG Stimulation for Crossover Study — Stimulation will be delivered on the left angular cortex (AG) using a real coil for 20 minutes with a frequency of 20Hz (train duration: 4s; inter-train interval: 26s; 3200 pulses at 80% of the resting motor threshold ) in one session. A single session will be conducted.
  Arms: AG Stimulation Group for Crossover Study
Device: Sham Stimulation for Parallel Study — Stimulation will be delivered on the dorsolateral prefrontal cortex (DLPFC) or the angular cortex (AG) using a sham coil for 20 minutes with a frequency of 20Hz (train duration: 4s; inter-train interval: 26s; 3200 pulses at 80% of the resting motor threshold ) in one session. Twenty sessions will be conducted.
  Arms: Sham Stimulation Group for Parallel Study (DLPFC + AG)
Device: DLPFC Stimulation for Parallel Study — Stimulation will be delivered on the left dorsolateral prefrontal cortex (DLPFC) using a real coil for 20 minutes with a frequency of 20Hz (train duration: 4s; inter-train interval: 26s; 3200 pulses at 80% of the resting motor threshold ) in one session. Twenty sessions will be conducted.
  Arms: DLPFC Stimulation Group for Parallel Study
Device: AG Stimulation for Parallel Study — Stimulation will be delivered on the left angular cortex (AG) using a real coil for 20 minutes with a frequency of 20Hz (train duration: 4s; inter-train interval: 26s; 3200 pulses at 80% of the resting motor threshold ) in one session. Twenty sessions will be conducted.
  Arms: AG Stimulation Group for Parallel Study

SUMMARY:
Background:

Severe brain injury could cause chronic disorders of consciousness (DOC). Treating DOC patients to improve recovery remains very challenging. A few randomized controlled studies have been published in the recent years, focusing on non-invasive brain stimulation (NIBS) treatments to improve patients' neurobehavioural functioning. Among NIBS, repetitive transcranial magnetic stimulation (rTMS) is a non-invasive brain stimulation technique that can modulate cortical excitability, enhance neural plasticity, and induce strong neuromodulatory effects that outlast the period of stimulation. It is thought to modulate cortical activity and could therefore be effective for treating DOC patients. Currently, there is no unified protocol for rTMS in DOC patients and studies vary in many aspects.

In this study, the investigators aim to improve the functional recovery of DOC patients following severe brain injury using rTMS in two multi-center double-blind studies.

Methods/design:

The investigators will recruit 90 DOC patients. Patients will have three rTMS sessions that will be randomized within patients in a crossover design: (i) one real stimulation on the left dorsolateral prefrontal cortex (DLPFC); (ii) one real stimulation on the left angular cortex (AG) and (iii) one sham stimulation. Sessions will be separated by at least 5 days washout period. Each stimulation session will last 20 minutes with a frequency of 20Hz (train duration: 4s; inter-train interval: 26s; 3200 pulses at 80% of the resting motor threshold - RMT). The RMT, i.e., the minimum stimulus intensity that generated a motor evoked potential response of at least 50μV at rest for 5 out of 10 trials, will be calculated for the stimulation target using single-pulses on the right abductor pollicis brevis muscle.

After an interval of one week, a parallel design study will begin. Ninety patients will be randomly divided in two experimental groups and one sham group (30 patients per group). Stimulation will be performed for 20 working days once a day with the same stimulation parameters as in the crossover study.

Primary outcome will be determined as behavioral response to treatment as measured using the Coma Recovery Scale - Revised (CRS-R). Resting-state high-density EEG will be also recorded to investigate the neurophysiological correlates by rTMS.

Discussion:

This study will contribute to define the role of rTMS for the treatment of DOC patients and characterise the neural correlates of its action. In addition, the investigators will define the responders' profile based on patients' characteristics and functional impairments and develop biomarkers of responsiveness using machine learning to categorize EEG signals according to clinical responsiveness to the treatment.

ELIGIBILITY:
Inclusion Criteria:

* over 18 years old
* > 28 days post-injury
* patients with DOC due to acquired brain lesions classified according to international guidelines as UWS or MCS with repeated behavioural assessments with the CRS-R
* stable vital parameters
* no previous neurological deficits anterior to the brain lesions
* no pregnancy
* no contraindication for rTMS or EEG (e.g., uncontrolled epilepsy, that is, seizure within 4 weeks prior to enrollment, metallic implant in the skull, pacemaker, craniotomy under the stimulated site, implanted brain device, sensitive skin)
* no sedative drugs and drugs thought to interfere with brain stimulation such as Na or Ca channel blockers (e.g., carbamazepine) or NMDA receptor antagonists (e.g., dextromethorphan)
* no drugs or substances which have strong potential of seizure induction (imipramine, amitriptyline, doxepin, nortriptyline, maprotiline, chlorpromazine, clozapine, foscarnet, ganciclovir, ritonavir, amphetamines, cocaine, phencyclidine, ketamine, gamma-hydroxybutyrate, alcohol, and theophylline).
* All etiologies (e.g., trauma, stroke, and anoxia)

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2024-07 (Estimated); Primary Completion 2024-11 (Estimated); Study Completion 2025-01 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline Coma Recovery Scale - Revised for Crossover Study | immediately after each rTMS session
  The Coma Recovery Scale - Revised is a non-invasive behavioural examination. It contains 23 items hierarchically presented and divided in 6 sub-scales (auditory, visual, motor, oro-motor/verbal, communication and arousal). The score is based on presence or absence of behaviours in response to sensory stimulations. The quantitative score can be calculated by adding the best observed response in each sub-scale. The diagnosis is obtained from the quality of observed behaviours (e.g., the ability of visual tracking means that the patient is minimally conscious). The total score ranges between 0 and 23. Higher scores mean a better outcome.
Change from Baseline Coma Recovery Scale - Revised for Parallel Study 1 | immediately after the last rTMS session
  The Coma Recovery Scale - Revised is a non-invasive behavioural examination. It contains 23 items hierarchically presented and divided in 6 sub-scales (auditory, visual, motor, oro-motor/verbal, communication and arousal). The score is based on presence or absence of behaviours in response to sensory stimulations. The quantitative score can be calculated by adding the best observed response in each sub-scale. The diagnosis is obtained from the quality of observed behaviours (e.g., the ability of visual tracking means that the patient is minimally conscious). The total score ranges between 0 and 23. Higher scores mean a better outcome.
Change from Baseline Coma Recovery Scale - Revised for Parallel Study 2 | 1 week after the last rTMS session
  The Coma Recovery Scale - Revised is a non-invasive behavioural examination. It contains 23 items hierarchically presented and divided in 6 sub-scales (auditory, visual, motor, oro-motor/verbal, communication and arousal). The score is based on presence or absence of behaviours in response to sensory stimulations. The quantitative score can be calculated by adding the best observed response in each sub-scale. The diagnosis is obtained from the quality of observed behaviours (e.g., the ability of visual tracking means that the patient is minimally conscious). The total score ranges between 0 and 23. Higher scores mean a better outcome.
Change from Baseline Coma Recovery Scale - Revised for Parallel Study 3 | 2 week after the last rTMS session
  The Coma Recovery Scale - Revised is a non-invasive behavioural examination. It contains 23 items hierarchically presented and divided in 6 sub-scales (auditory, visual, motor, oro-motor/verbal, communication and arousal). The score is based on presence or absence of behaviours in response to sensory stimulations. The quantitative score can be calculated by adding the best observed response in each sub-scale. The diagnosis is obtained from the quality of observed behaviours (e.g., the ability of visual tracking means that the patient is minimally conscious). The total score ranges between 0 and 23. Higher scores mean a better outcome.

SECONDARY OUTCOMES:
Change from Baseline Resting-State EEG for Crossover Study 1 | during each rTMS session
  EEG will be collected using a high-density EEG. Fifteen minutes of resting state will be performed. Resting-state EEG complexity and connectivity analyses will be performed at the individual and group level. The investigators will compute spectral measures as well as cortical functional connectivity using median spectral connectivity and graph-theoretic topology metrics such as clustering coefficient, path length, modularity and participation coefficient.
Change from Baseline Resting-State EEG for Crossover Study 2 | immediately after each rTMS session
  EEG will be collected using a high-density EEG. Fifteen minutes of resting state will be performed. Resting-state EEG complexity and connectivity analyses will be performed at the individual and group level. The investigators will compute spectral measures as well as cortical functional connectivity using median spectral connectivity and graph-theoretic topology metrics such as clustering coefficient, path length, modularity and participation coefficient.
Change from Baseline Resting-State EEG for Parallel Study 1 | immediately after the last rTMS session
  EEG will be collected using a high-density EEG. Fifteen minutes of resting state will be performed. Resting-state EEG complexity and connectivity analyses will be performed at the individual and group level. The investigators will compute spectral measures as well as cortical functional connectivity using median spectral connectivity and graph-theoretic topology metrics such as clustering coefficient, path length, modularity and participation coefficient.
Change from Baseline Resting-State EEG for Parallel Study 2 | 1 week after the last rTMS session
  EEG will be collected using a high-density EEG. Fifteen minutes of resting state will be performed. Resting-state EEG complexity and connectivity analyses will be performed at the individual and group level. The investigators will compute spectral measures as well as cortical functional connectivity using median spectral connectivity and graph-theoretic topology metrics such as clustering coefficient, path length, modularity and participation coefficient.
Change from Baseline Resting-State EEG for Parallel Study 3 | 2 week after the last rTMS session
  EEG will be collected using a high-density EEG. Fifteen minutes of resting state will be performed. Resting-state EEG complexity and connectivity analyses will be performed at the individual and group level. The investigators will compute spectral measures as well as cortical functional connectivity using median spectral connectivity and graph-theoretic topology metrics such as clustering coefficient, path length, modularity and participation coefficient.

CONTACTS AND LOCATIONS:
Locations (2):
- University Hospital of Liège, Liège, Belgium
- Therapiezentrum Burgau, Burgau, Germany

REFERENCES:
- [Derived] Vitello MM, Rosenfelder MJ, Cardone P, Niimi M, Willacker L, Thibaut A, Lejeune N, Laureys S, Bender A, Gosseries O. A protocol for a multicenter randomized and personalized controlled trial using rTMS in patients with disorders of consciousness. Front Neurol. 2023 Jul 21;14:1216468. doi: 10.3389/fneur.2023.1216468. eCollection 2023. PMID 37545735